CLINICAL TRIAL: NCT03056872
Title: Physiological Stress Reactivity as a Determinant in Co-occurring Alcohol Use and Anxiety Disorder: Diagnosis and Alcohol Use Outcomes
Brief Title: Stress Reactivity as a Determinant in Co-occurring Alcohol Use and Anxiety Disorder: Diagnosis and Alcohol Use Outcomes
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: PSYCH-2017-23713; 1K01AA024805 (NIH)
Record Dates: First submitted 2017-02-09; First posted 2017-02-17 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder; Anxiety Disorder/Anxiety State; Stress Disorder; Hypothalamic Pituitary Adrenal; Drinking to Cope
MeSH Terms: conditions — Alcoholism; Anxiety Disorders; Stress Disorders, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AUD only: AUD treatment inpatients without a co-occurring AnxD receiving AUD treatment as usual
- AnxD+AUD-Cognitive Behavioral Therapy (CBT): AUD treatment inpatients with a co-occurring anxiety disorder receiving AUD treatment as usual in addition to CBT for co-occurring AUD+AnxD
- AnxD+AUD- No CBT: AUD treatment inpatients with a co-occurring anxiety disorder receiving AUD treatment as usual only.
- Healthy Controls: Community sample

SUMMARY:
Alcohol dependence is among the most common and costly public health problems affecting the nation. Among individuals with alcohol use disorder (AUD), those with (vs. without) a co-occurring anxiety disorder (AnxD) are as much as twice as likely to relapse in the months following AUD treatment. Dysregulation of biological stress-mood systems predict and correlate with AUD relapse and AnxD symptomatology. In contrast, stress system re-regulation correlates with improved AUD treatment outcomes but has not been examined with respect to AUD recovery and relapse in co-occurring AUD+AnxD.

DETAILED DESCRIPTION:
The objectives of the proposed research are to 1) evaluate the effect of co-occurring AnxD on the severity of biological stress-mood system dysregulations in AUD inpatients at pre-treatment, 2) evaluate the effect of co-occurring AnxD on the persistence of stress-mood system dysregulations in AUD inpatients in the months following treatment, 3) evaluate the effects of treatment on biological stress-mood system re-regulation among AUD patients with co-occurring AnxD, and 4) evaluate the effect of re-regulation change in biological stress-mood system function on AUD clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Between the ages of 18 and 65
* Diagnostic and Statistical Manual diagnosis of a Panic Disorder, Generalized Anxiety Disorder, or Social Anxiety Disorder within the past 30 days (AUD+AnxD group only).
* Primary alcohol use disorder diagnosis and alcohol use in the 30 days preceding the study (AUD alone and AUD+AnxD groups only).
* Inpatient treatment at Lodging Plus primarily for alcohol (vs. other drug with nicotine accepted) dependence (AUD alone and AUD+AnxD groups only).
* A minimum of a sixth-grade reading level.
* Healthy controls, same criteria absent AUD and AnxD diagnosis of an alcohol and/or anxiety disorder
* Lives within proximity to the Twin Cities (e.g., within about an hour's drive) or willing to drive to Fairview for the purpose of attending follow-up visits
* Willingness to provide contact information to confirm follow-up appointments

Exclusion Criteria:

* Lifetime history of psychosis or mania
* Cognitive impairment, physical impairment, or chronic medical illness that precludes study participation
* Primary PTSD as determined by qualifying assessment
* Females currently pregnant
* Exposure to antipsychotic medication for a total duration >16 weeks.
* Prior head injury leading to >30 minutes of unconsciousness.
* Cognitive impairment that impedes study participation.
* Healthy controls with a history of any major medical or psychiatric disorders (e.g., schizophrenia, depression, heart disease, or stroke).
* Suicide intent or attempt in the past 30 days
* Cardiovascular health issues
* Thyroid Disease
* History of severe neurological illness such as chronic seizure disorder (e.g, epilepsy) or stroke
* Brain tumor and/or implants in the skull cavity (e.g., plate in the skull)
* Pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 1) inpatients receiving treatment for an alcohol use disorder 2) healthy controls recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Relapse Status | 4-month follow-up
  Relapse status will be assessed using a categorical measure of whether someone did vs did not drink (yes vs. no) during the 4 months following treatment discharge.
Relapse Severity | 4-month follow-up
  Relapse severity will consist of the number days drinking during the 4 months following treatment discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Anker, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Fairview Riverside, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No